CLINICAL TRIAL: NCT02007135
Title: Comparison of fMRI Compatible Pneumatic and Electromagnetic Muscle Vibrators to Stimulate Muscle Proprioceptors
Brief Title: Comparison of Pneumatic and Electromagnetic Muscle Vibrators to Stimulate Muscle Proprioceptors
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Simon Brumagne, Professor Simon Brumagne, KU Leuven
Other Study IDs: 2013_SBrumagne_pneumvibrators
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Proprioceptive Postural Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy: Healthy persons, without non-specific low back pain

SUMMARY:
The purpose of this study is to determine the concurrent validity of a newly developed pneumatic, fMRI compatible muscle vibrator as compared to a electromagnetic muscle vibrator in the stimulation of muscle proprioceptors.

ELIGIBILITY:
Inclusion criteria for healthy individuals:

* Age: 20-45 years old
* No history of low back pain
* A score of 0% on the Oswestry Disability Index
* Willingness to sign the informed consent

Exclusion Criteria:

* History of major trauma and/or major orthopedic surgery of the spine, pelvis or lower quadrant
* One of the following conditions: Parkinson, MS, Stroke with sequels....
* Radicular symptoms
* Not Dutch-speaking
* Strong opioids
* Neck pain
* Ankle problems
* Smoking

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young Flemish Volunteers
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Proprioceptive postural control | 6 months
  Center of pressure displacement on a force plate in standing in response to local muscle vibration on ankle and back muscles to specifically detect the role of proprioception in postural control.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brumagne, Professor, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

REFERENCES:
- [Background] Claeys K, Brumagne S, Dankaerts W, Kiers H, Janssens L. Decreased variability in postural control strategies in young people with non-specific low back pain is associated with altered proprioceptive reweighting. Eur J Appl Physiol. 2011 Jan;111(1):115-23. doi: 10.1007/s00421-010-1637-x. Epub 2010 Sep 8. PMID 20824281